TR Istanbul University-Cerrahpaşa ID: İstanbul UCEdu

Informed Consent Form: June 1, 2023
The effect of two different bathing methods on vital parameters and stress levels in preterm babies.

Clinical Trial Number: NCT06166485

## TR Istanbul University-Cerrahpaşa

## Social and Humanities Research Ethics Committee

## INFORMED VOLUNTARY CONSENT FORM

You Prof. Dr. Under the supervision of Sevil İnal, Prof. Dr. Sevil İnal and Midwife Ayşe Dilan Koçak "The effect of bathing applied in two different orders on the stress level and physiological parameters in term babies" conducted by We invite you to the research titled. The aim of this study is to determine the effect of bathing applied in two different orders (first the body and then the head, and the classical method of washing the whole body, starting from the head) on the stress level and physiological parameters in healthy babies born at term . Scales/interview forms/data collection tools called Newborn Stress Scale will be used in the research . You are expected to spend approximately 30 minutes for the research. 104 people, including your baby, will participate in the research. Participating in this study is entirely voluntary. In order to achieve the purpose of the study, what is expected from you is to answer sincerely and give the answers that best suit you, without being under anyone's pressure or suggestion. Reading and approving this form will mean that you agree to participate in the research. However, not participating in the study or withdrawing from the study at any time after participating You have the right. The information obtained from this study will be used entirely for research purposes and your personal information will be kept confidential; However, your data may be used for publication purposes. Your contact information can only be transferred to the "common participant pool" with your permission and so that different researchers can contact you. All data collected in the research will be kept completely confidential and will not be shared with anyone outside the research team. Data stored digitally will be protected by encryption method; Data on paper will be kept in a locked cabinet. All collected data will be irreversibly destroyed within 2 years after the completion of the study. If you need more information now or later, apart from the information given about the purpose of the research, you can ask the researcher now or contact the researcher via e-mail address inalsevil@gmail.com and phone number 05334332824. If you would like general/specific results to be shared with you when the research is completed, please notify the researcher.

Information if audio and video recording will be made: Audio and video recording will not be made.

data will be collected online: Data will be collected while performing the application.

I have read the above information that should be given to the participant before the research, and I understand the scope and purpose of the study in which I am asked to participate and my responsibilities as a volunteer. Written and verbal explanations about the study were made by the researcher/researchers named below. The possible risks and benefits of the study were also explained to me verbally. I was given sufficient confidence that my personal information would be carefully protected.

Under these circumstances. I conducted the research in question voluntarily, without any pressure or

| onder these enganistances, I conducted the research in question voluntarity, without any pressure of |
|---|
| suggestion. I agree to participate without |
| Participant: |
| Name-Surname: |
| Signature: Contact Information: e-mail: Phone: |
| Transferring my contact information to the "common research pool" so that other researchers can contact me; $\Box$ I |
| accept $\Box$ I do not accept (please select the appropriate option) |
| For Those Under Guardianship or Guardianship; |
| Name-Surname of Parent or Guardian: |
| Signature: |

of the researcher

